

| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Version Number: | 3.1 |
| | Effective Date: | 25-Nov-2021 |

# Statistical Analysis Plan

# Study Title

A Postmarketing, Phase 4, Multicentre, Prospective, Single- arm study to Assess the Safety of Fasenra® (Benralizumab) in Adult Patients of Severe Asthma with Eosinophilic Phenotype in India

| ( 'X' | | |
|---|---|---|
| Protocol/ Study Number | : | D3250C00093 |
| Sponsor Name | : | AstraZeneca Pharma India Limited |
| Sponsor Address | | AstraZeneca Pharma India Limited,<br>Block N1, 12th Floor, Manyata Embassy Business<br>Park<br>Rachenahalli, Outer Ring Road, Bangalore-560045 |
| Document Version | | 1.1 |
| Document Date | : / | 12-Jun-2024 |
| Author Name (s) | : | PPD |
| Designation | : | PPD |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Version Number: | 3.1 | |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# **Table of Contents**

| LIST OF TABLE | |
|--------------------------------------------------------|--------------|
| LIST OF LISTING | 8 |
| LIST OF FIGURES | 10 |
| LIST OF ABBREVIATION | 11 |
| 1. INTRODUCTION | 12 |
| 2. Study Objective and Design | 12 |
| 2.1 Study Objective | 12 |
| 2.1.1 Primary Objective | 12 |
| 2.1.2 Secondary Objective | 12 |
| 2.2 Study Description | 12 |
| 2.2.1 Study Design | 12 |
| 2.2.2 Inclusion Criteria | 13 |
| 2.2.3 Exclusion Criteria | 14 |
| 2.2.4 Study Flow chart | 15 |
| 2.2.5 Study Plan | 16 |
| 2.3 Randomization | 17 |
| 2.4 Blinding and Un-Blinding | 17 |
| 2.5 Interim Analysis | 17 |
| 3. Population Analysis Set | 17 |
| 3.1 Enrolled Analysis Set | 17 |
| 3.2 Assigned to Study intervention Analysis Set | 17 |
| 3.3 Evaluable Analysis Set | 17 |
| 3.4 Safety Analysis Set | 17 |
| 4. Sample Size and Power Calculations | 17 |
| 5. Patient Characteristics and Study Conduct Summaries | 18 |
| 5.1 General Considerations | 18 |
| 5.2 Decimal Point | 18 |
| 5.3 Disposition of Patients | 18 |
| 5.4 Demographic and Baseline Characteristics | 19 |
| 5.5 Covid-19 Vaccination | 19 |
| 5.6 Medical History | 19 |
| 5.7 Electrocardiogram (ECG) | 19 |
| Document | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| 6. Endpoints Analysis Strategy | 20 |
|---|---|
| 6.1 Endpoints Analysis | 20 |
| 6.1.1 Primary Endpoint | 20 |
| 6.1.2 Secondary Endpoint | 20 |
| 6.2 Efficacy Hypothesis | 20 |
| 6.3 Statstical Methods for Efficacy Analsysis | 20 |
| 6.3.1 Primary Endpoint Analysis | 20 |
| 6.3.2 Secondary Endpoint Analysis | 22 |
| 7. References | 23 |
| 8. Mock Tables | 24 |
| Table 14.1.1.1. Patient Disposition in the Study (Enrolled Analysis Set) | 24 |
| Table 14.1.1.2. Summary of Patient Discontinuation of Study Intervention (Evaluable Analysis Set ) | 25 |
| Table 14.1.1.3. Summary of Analysis Population (Enrolled Analysis Set) | 26 |
| Table 14.1.2.1. Summary of Demographic and Baseline Characteristics (Evaluable Analysis Set) | 26 |
| Table 14.1.2.2. Summary of Anthropometric Assessment (Evaluable Analysis Set) | 27 |
| Table 14.1.3. Summary of Significant Medical History (Evaluable Analysis Set) | 28 |
| Table 14.1.4. Summary of COVID-19 vaccination (Evaluable Analysis Set) | 29 |
| Table 14.1.5.1. Summary of Prior Asthma Therapy (Evaluable Analysis Set) | 30 |
| Table 14.1.5.2. Summary of oral/inhaled Corticosteroid (Evaluable Analysis Set) | 31 |
| Table 14.1.6. Patient Administration of Benralizumab (Evaluable Analysis Set) | 32 |
| Table 14.1.7. Summary of Overdose (Evaluable Analysis Set) | 33 |
| Table 14.1.8. Summary of Pulmonary Function Test (Evaluable Analysis Set) | 34 |
| Table 14.2.1.1. Summary of Asthma and Exacerbation (Evaluable Analysis Set) | 36 |
| Table 14.2.1.2. Summary of Exacerbation (Evaluable Analysis Set) | 37 |
| Table 14.2.1.3. Summary of Before and After Treatment Exacerbation (Evaluable Analysis Set) | 38 |
| Table 14.2.2. Summary of Time to first Exacerbation (Evaluable Analysis Set) | 39 |
| Table 14.2.3. Analysis of change in Blood Eosinophils count from baseline to Visit 2, Visit 4 and Visit 5 (Eva | |
| Table 14.2.4 Summary of Overall Investigators Assessment (Evaluable Analysis Set) | 41 |
| Table 14.3.1.1. Overall Summary of Adverse Events (Safety Analysis Set) | 42 |
| Table 14.3.1.2. Summary of Treatment Emergent Adverse Events (Safety Analysis Set) | 43 |
| Table 14.3.1.3.1 Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred T Analysis Set) | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Document Page 4 of 9 | )5 |
|---|---|
| Listing 16.2.3. Listing of Patient Blood Eosinophils count | 76 |
| Listing 16.2.2.3. Listing of Patient Exacerbation (Part 3) | 75 |
| Listing 16.2.2.2. Listing of Patient Exacerbation (Part 2) | 74 |
| Listing 16.2.2.1. Listing of Patient Exacerbation (Part 1) | 73 |
| Listing 16.2.1.2. Listing of Patient Assessment of Asthma and Exacerbation | 72 |
| Listing 16.2.1.1. Listing of Patient Asthma and Exacerbation History | 71 |
| Listing 16.1.7. Listing of Patient Pulmonary Function Test | 70 |
| Listing 16.1.6.2. Listing of Patient Overdose | 69 |
| Listing 16.1.6.1. Listing of Patient Administration of Benralizumab | 68 |
| Listing 16.1.5.2. Listing of Patient Prior Oral/Inhaled Corticosteroid Therapy | 67 |
| Listing 16.1.5.1. Listing of Patient Prior Asthma Therapy | 66 |
| Listing 16.1.4. Listing of Patient COVID-19 Vaccination | 65 |
| Listing 16.1.3. Listing of Patient Significant Medical History | 64 |
| Listing 16.1.2.2. Listing of Patient Anthropometry | 63 |
| Listing 16.1.2.1. Listing of Patient Demographics Information | 62 |
| Listing 16.1.1.4. Listing of Patient Analysis Set | 61 |
| Listing 16.1.1.3. Listing of Patient Study Completion | 60 |
| Listing 16.1.1.2. Listing of Patient Discontinuation of Study Intervention | 59 |
| Listing 16.1.1.1. Listing of Patient Informed consent | 58 |
| Table 14.3.6.2. Summary of Urine Pregnancy Test (Safety Analysis Set) | 57 |
| Table 14.3.6.1. Summary of Serum Pregnancy Test (Safety Analysis Set) | 56 |
| Table 14.3.5. Summary of Targeted Physical Examination (Safety Analysis Set) | 54 |
| Table 14.3.4. Summary of Electrocardiogram (Safety Analysis Set) | 52 |
| Table 14.3.3. Analysis of change in Vital Sign parameters from baseline to Visit 1, Visit 2, Visit 3, Visit 4 and Vi<br>(Safety Analysis Set) | |
| Table 14.3.2.2. Analysis of change in Biochemistry parameters from baseline to Week 24 (Safety Analysis Set) | ) 50 |
| Table 14.3.2.1. Analysis of change in Haematology parameters from baseline to Week 24. (Safety Analysis Set | t)49 |
| Table 14.3.1.6. Summary of Serious TEAE by System Organ Class and Preferred Term (Safety Analysis Set) | |
| Table 14.3.1.5. Summary of TEAE leading to discontinuation by System Organ Class and Preferred Term (Safe<br>Analysis Set) | • |
| Table 14.3.1.4. Summary of TEAE related to the Investigational Product by System Organ Class and Preferred (Safety Analysis Set) | |
| (Safety Analysis Set) | 45 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Listing 16.2.4. Listing of Overall Investigators Assessment | 77 |
|-----------------------------------------------------------------------|----|
| Listing 16.3.1.1. Listing of Patient Adverse Event Assessment | 78 |
| Listing 16.3.1.2. Listing of Patient Adverse Events | 79 |
| Listing 16.3.2.1. Listing of Patient Serious Adverse Events (Part 1) | 80 |
| Listing 16.3.2.2. Listing of Patient Serious Adverse Events (Part 2) | 81 |
| Listing 16.3.3.1. Listing of Patient Haematology Parameters | 82 |
| Listing 16.3.3.2. Listing of Patient Biochemistry Parameters | 83 |
| Listing 16.3.3. Listing of Patient Urinalysis Parameters | 84 |
| Listing 16.3.3.4. Listing of Patient Serum Pregnancy Test | 85 |
| Listing 16.3.4. Listing of Patient Vital Signs | 86 |
| Listing 16.3.5. Listing of Patient Electrocardiogram (ECG) | 87 |
| Listing 16.3.6. Listing of Patient Targeted Physical Examination | 88 |
| Listing 16.3.7. Listing of Patient Urinalysis Pregnancy test | 89 |
| Listing 16.3.8. Listing of Patient Pregnancy Form | 90 |
| Listing 16.3.9.1. Listing of Patient Concomitant Medication | 91 |
| Listing 16.3.9.2. Listing of Patient Prior and Concomitant Medication | 92 |
| Figure 14.2.1. Figure of Time to first Asthma Exacerbation | 93 |
| Figure 14.2.2. Figure of Number of Exacerbation | 94 |
| Figure 14.2.3. Figure of Mean of Exacerbation | 95 |



| | Document Title: | Document ID: | BP04-01 |
|---|---|---|---|
| Canadination Appril 1910 Plant | Version Number: | 3.1 | |
| | Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# LIST OF TABLE

| Table 14.1.1.1. Patient Disposition in the Study (Enrolled Analysis Set) | 24 |
|---|---|
| Table 14.1.1.2. Summary of Patient Discontinuation of Study Intervention (Evaluable Analysis Set ) | 25 |
| Table 14.1.1.3. Summary of Analysis Population (Enrolled Analysis Set) | 26 |
| Table 14.1.2.1. Summary of Demographic and Baseline Characteristics (Evaluable Analysis Set) | |
| Table 14.1.2.2. Summary of Anthropometric Assessment (Evaluable Analysis Set) | 27 |
| Table 14.1.3. Summary of Significant Medical History (Evaluable Analysis Set) | 28 |
| Table 14.1.4. Summary of COVID-19 vaccination (Evaluable Analysis Set) | 29 |
| Table 14.1.5.1. Summary of Prior Asthma Therapy (Evaluable Analysis Set) | |
| Table 14.1.5.2. Summary of oral/inhaled Corticosteroid (Evaluable Analysis Set) | |
| Table 14.1.6. Patient Administration of Benralizumab (Evaluable Analysis Set) | 32 |
| Table 14.1.7. Summary of Overdose (Evaluable Analysis Set) | 33 |
| Table 14.1.8. Summary of Pulmonary Function Test (Evaluable Analysis Set) | |
| Table 14.2.1.1. Summary of Asthma and Exacerbation (Evaluable Analysis Set) | 36 |
| Table 14.2.1.2. Summary of Exacerbation (Evaluable Analysis Set) | |
| Table 14.2.1.3. Summary of Before and After Treatment Exacerbation (Evaluable Analysis Set) | |
| Table 14.2.2. Summary of Time to first Exacerbation (Evaluable Analysis Set) | 39 |
| Table 14.2.3. Analysis of change in Blood Eosinophils count from baseline to Visit 2, Visit 4 and Visit 5 (Evaluable | |
| Analysis Set) | 40 |
| Table 14.2.4 Summary of Overall Investigators Assessment (Evaluable Analysis Set) | |
| Table 14.3.1.1. Overall Summary of Adverse Events (Safety Analysis Set) | 42 |
| Table 14.3.1.2. Summary of Treatment Emergent Adverse Events (Safety Analysis Set) | 43 |
| Table 14.3.1.3.1 Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Sai | |
| Analysis Set) | |
| <u>Table 14.3.1.3.2 Summary of Serious Treatment Emergent Adverse Events by System Organ Class and Preferred To</u> (Safety Analysis Set) | |
| Table 14.3.1.4. Summary of TEAE related to the Investigational Product by System Organ Class and Preferred Tern | |
| (Safety Analysis Set) | |
| Table 14.3.1.5. Summary of TEAE leading to discontinuation by System Organ Class and Preferred Term (Safety | |
| Analysis Set) | 47 |
| Table 14.3.1.6. Summary of Serious TEAE by System Organ Class and Preferred Term (Safety Analysis Set) | 48 |
| Table 14.3.2.1. Analysis of change in Haematology parameters from baseline to Week 24. (Safety Analysis Set) | 49 |
| Table 14.3.2.2. Analysis of change in Biochemistry parameters from baseline to Week 24 (Safety Analysis Set) | 50 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Table 14.3.3. Analysis of change in Vital Sign parameters from baseline to Visit 1, Visit 2, Visit 3, Visit 4 and Visit 5 | |
|---|---|
| (Safety Analysis Set) | .51 |
| Table 14.3.4. Summary of Electrocardiogram (Safety Analysis Set) | . 52 |
| Table 14.3.5. Summary of Targeted Physical Examination (Safety Analysis Set) | .54 |
| Table 14.3.6.1. Summary of Serum Pregnancy Test (Safety Analysis Set) | |
| Table 14.3.6.2. Summary of Urine Pregnancy Test (Safety Analysis Set) | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# LIST OF LISTING

| <u>Listing 16.1.1.1. Listing of Patient Informed consent</u> | 58 |
|---|---|
| Listing 16.1.1.2. Listing of Patient Discontinuation of Study Intervention | |
| Listing 16.1.1.3. Listing of Patient Study Completion | 60 |
| Listing 16.1.1.4. Listing of Patient Analysis Set | 61 |
| Listing 16.1.2.1. Listing of Patient Demographics Information | 62 |
| Listing 16.1.2.2. Listing of Patient Anthropometry | 63 |
| Listing 16.1.3. Listing of Patient Significant Medical History | 64 |
| Listing 16.1.4. Listing of Patient COVID-19 Vaccination | 65 |
| Listing 16.1.5.1. Listing of Patient Prior Asthma Therapy | 66 |
| Listing 16.1.5.2. Listing of Patient Prior Oral/Inhaled Corticosteroid Therapy | 67 |
| Listing 16.1.6.1. Listing of Patient Administration of Benralizumab | 68 |
| Listing 16.1.6.2. Listing of Patient Overdose | 69 |
| Listing 16.1.7. Listing of Patient Pulmonary Function Test | 70 |
| Listing 16.2.1.1. Listing of Patient Asthma and Exacerbation History | 71 |
| Listing 16.2.1.2. Listing of Patient Assessment of Asthma and Exacerbation | 72 |
| Listing 16.2.2.1. Listing of Patient Exacerbation (Part 1) | 73 |
| Listing 16.2.2.2. Listing of Patient Exacerbation (Part 2) | 74 |
| Listing 16.2.2.3. Listing of Patient Exacerbation (Part 3) | 75 |
| Listing 16.2.3. Listing of Patient Blood Eosinophils count | 76 |
| Listing 16.2.4. Listing of Overall Investigators Assessment | 77 |
| Listing 16.3.1.1. Listing of Patient Adverse Event Assessment | 78 |
| Listing 16.3.1.2. Listing of Patient Adverse Events | 79 |
| Listing 16.3.2.1. Listing of Patient Serious Adverse Events (Part 1) | 80 |
| Listing 16.3.2.2. Listing of Patient Serious Adverse Events (Part 2) | 81 |
| Listing 16.3.3.1. Listing of Patient Haematology Parameters | 82 |
| Listing 16.3.3.2. Listing of Patient Biochemistry Parameters | 83 |
| Listing 16.3.3.3. Listing of Patient Urinalysis Parameters | 84 |
| Listing 16.3.3.4. Listing of Patient Serum Pregnancy Test | 85 |
| Listing 16.3.4. Listing of Patient Vital Signs | 86 |
| Listing 16.3.5. Listing of Patient Electrocardiogram (ECG) | 87 |
| Listing 16.3.6. Listing of Patient Targeted Physical Examination | 88 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Listing 16.3.7. Listing of Patient Urinalysis Pregnancy test | 89 |
|-----------------------------------------------------------------------|----|
| Listing 16.3.8. Listing of Patient Pregnancy Form | 90 |
| Listing 16.3.9.1. Listing of Patient Concomitant Medication | 91 |
| Listing 16.3.9.2. Listing of Patient Prior and Concomitant Medication | 92 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# LIST OF FIGURES

| Figure 14.2.1. Figure of Time to first Asthma Exacerbation | .93 |
|------------------------------------------------------------|-----|
| Figure 14.2.2. Figure of Number of Exacerbation | .94 |
| Figure 14.2.3. Figure of Mean of Exacerbation. | .95 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# LIST OF ABBREVIATION

| Abbreviation | Term |
|--------------|-----------------------------------------|
| ADA | antidrug antibody |
| ADR | adverse drug reaction |
| AE | adverse event |
| CI | confidence interval |
| COPD | chronic obstructive pulmonary disease |
| CRO | contract research organisation |
| ECG | electrocardiogram |
| EDC | electronic data capture |
| ER | Emergency Room |
| eCRF | electronic case report form |
| EOS | End of Study |
| FEV1 | forced expiratory volume in 1 second |
| GCP | Good Clinical Practice |
| GINA | Global Initiative for Asthma |
| ICS | inhaled corticosteroid |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IL-5 | interleukin-5 |
| IL-5Rα | interleukin-5 receptor alpha subunit |
| IMP | Investigational Medicinal Product |
| IRB | Institutional Review Board |
| KM | Kaplan-Meier |
| LABA | long-acting beta-agonist |
| OCS | 8.1.Oral corticosteroid |
| PI | Package Insert |
| Pre-BD | prebronchodilator |
| Post-BD | postbronchodilator |
| SAE | serious adverse event |
| SD | standard deviation |
| SAP | statistical analysis plan |
| SmPC | Summary of product characteristics |
| SoA | schedule of activities |
| TEAE | treatment-emergent adverse event |
| USPI | United States Prescribing Information |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

#### 1. INTRODUCTION

The purpose of this document is to provide a description of the statistical methods and procedures to be implemented for the analysis of data from D3250C00093 study. This document is based on protocol V 1.0, 09 Mar 2021. The statistical planning and conduct of analysis of the data from this study will follow the principles defined in relevant International Council on Harmonisation (ICH)-E9 guidelines. Any change from the planned analysis as described in the protocol, are detailed here, and any differences described here supersede the analysis as presented in the protocol.

# 2. Study Objective and Design

### 2.1 Study Objective

#### 2.1.1 Primary Objective

 To Assess the safety and tolerability of Fasenra (Benralizumab) in adult patients of Severe asthma with eosinophilic phenotype over a period of 24 weeks.

#### 2.1.2 Secondary Objective

 To assess the effectiveness of Fasenra (benralizumab) in adult patients of severe asthma with eosinophilic phenotype over a period of 24 weeks

#### 2.2 Study Description

#### 2.2.1 Study Design

This is a Phase 4, single-arm, prospective, multicentre, interventional study, designed to assess the safety, tolerability, and effectiveness of benralizumab in adult patients of severe asthma with eosinophilic phenotype in India. The study is planned to meet the post approval commitment as a regulatory requirement.

Ten centres across India will participate in this study. The investigators will be pulmonologists or chest physicians treating asthma patients. Informed consent will be obtained from all the patients at screening before any study-related procedures are performed. Adult patients of severe asthma with eosinophilic phenotype, who are prescribed benralizumab as an add-on therapy by the treating physician, will be enrolled in the study.

The total study duration will be 24 weeks, including 16 weeks of study treatment, and 8 weeks follow-up.

- Screening duration: 2 weeks
- Study period: 24 weeks
- Treatment duration (4 doses): 16 weeks (Day 1, Week 4, Week 8, and Week 16)
- Post-treatment follow-up duration: 8 weeks (Week 24)

Participants will be maintained on their currently prescribed therapies including ICS-LABA therapy(ies), throughout the study duration.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Study population will include adult (18 to 75 years of age) male or female patients who have severe asthma with eosinophilic phenotype requiring high dose of ICS and LABA.

Each participant should meet all the inclusion criteria and none of the exclusion criteria to be eligible for the study.

Under no circumstances can there be exceptions to this rule. Participants who do not meet the entry requirements are screen failures

"Enrolled" means a participant's, or their legally acceptable representative's, agreement to participate in a clinical study after completion of the informed consent process. Prospective approval of protocol deviations to recruitment and enrolment criteria, also known as protocol waivers or exemptions, is not permitted.

This proposed Phase 4 single-arm study will fulfil the regulatory requirement as a postmarketing study to assess the safety of 30-mg benralizumab administered subcutaneously in Indian patients of severe asthma with eosinophilic phenotype who remain uncontrolled on high doses of ICS plus LABA. Owing to the recent marketing approval, there are no data available from real-life studies in the Indian population. Participants included in this study will be as per the indicated patient profile in the local prescribing information, specifically taking into consideration the contraindications, warnings, and special precautions for use.

The study will enrol patients who have been prescribed benralizumab as per the local prescribing information. The recommended dose is 30 mg administered once every 4 weeks for the first 3 doses, and then once every 8 weeks thereafter by subcutaneous injection into the upper arm, thigh, or abdomen by the study physician. Four doses of benralizumab will be administered as part of the study.

#### 2.2.2 Inclusion Criteria

Patients are eligible to be included in the study only if all of the following criteria apply:

- 1. Male or female patients 18 to 75 years of age inclusive, at the time of signing the informed consent
- 2. Patients with physician's confirmed diagnosis of severe asthma with an eosinophilic phenotype, ie, diagnosis of severe asthma in preceding at least 12 months, with an eosinophil count of ≥300 cells/μL at screening, requiring treatment with high-dose ICS (>500 μg fluticasone propionate dry powder formulation, or >800 μg budesonide dry powder formulation, or equivalent total daily dose) and a LABA as maintenance treatment for at least 3 months prior to enrolment
- A decreased lung function with prebronchodilator (Pre-BD) forced expiratory volume in 1 second (FEV1) of <80% predicted, demonstrated by spirometry at screening</li>
- 4. At least 2 documented asthma exacerbations in the preceeding12 months, except in 30 days before the date of informed consent, that required the use of a systemic corticosteroid or temporary increase from the patient's usual maintenance dose of OCS



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

- Documented postbronchodilator (post-BD) reversibility in FEV1 of ≥12% and ≥200 mL in FEV1 within 12
  months before first dose. If historical documentation is not available, reversibility must be demonstrated and
  documented at screening or Day 1 before first dose
- 6. Benralizumab naive patients who have not previously received benralizumab prior to the start of this study
- Patients who are willing and capable of giving signed informed consent as described in Appendix A, which
  includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in
  this protocol.

#### 2.2.3 Exclusion Criteria

Patients will be excluded from the study if any of the following criteria apply:

- Clinically important pulmonary disease other than asthma (eg, active lung infection, chronic obstructive
  pulmonary disease, bronchiectasis, pulmonary fibrosis, cystic fibrosis etc.) or ever been diagnosed with
  pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil
  counts (eg, allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic
  syndrome), which can confound the outcome assessment
- Patients currently enrolled in an interventional clinical study in parallel including those with any biologic treatment
- 3. Patients who have received any biologic within 30 days prior to the date of informed consent.
- Known history of allergy or reaction to the benralizumab formulation or excipients (L-histidine, L-histidine hydrochloride monohydrate, α-trehalose dihydrate, polysorbate 20, water for injection)
- 5. History of anaphylaxis to any biologic therapy
- A helminthic parasitic infection diagnosed within 24 weeks before the date informed consent is obtained that
  has not been treated with, or has failed to respond to, standard of care therapy
- 7. Acute asthma exacerbation 30 days before the date informed consent
- 8. Acute asthma exacerbation between screening and first dose of study dose administration.
- Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days before
  the date informed consent
- 10. Patients with malignancy within 5 years prior to enrolment, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal, or squamous cell carcinoma or non-melanomatous skin cancer with active or recent malignancy



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

- 11. Any clinically significant abnormal findings in physical examination, vital signs, haematology, clinical chemistry, or urinalysis, which, in the opinion of the investigator, may put the participant at risk because of his/her participation in the study
- 12. History of current alcohol, drug, or chemical abuse or past abuse that would impair or risk the participant's full participation in the study, in the opinion of the investigator
- 13. Female patients who are pregnant or lactating or planning a family during the study period.

# 2.2.4 Study Flow chart



EOS = end of study



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Die | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# 2.2.5 Study Plan

| | Screening | Intervention Period | | | Follow-up | |
|---|---|---|---|---|---|---|
| Procedure | (Up to 14 Days<br>Before Day 1) | Day 1 | Week 4 | Week 8 | (Last<br>Dose)Week 16 | EOS<br>Week 24 |
| | | | Day 28±2 | Day 56±2 | Day 112±2 | Day 168±7 |
| Visit | | 1 | 2 | 3 | 4 | 5 |
| Informed consent | X | | | | | |
| Inclusion and exclusion criteria* | X | | | | | |
| Demography, anthropometry including BMI | X | | | | | |
| Significant medical history | X | | | | | |
| Clinical safety laboratory assessments <sup>b</sup> | X | | | | | X |
| Serum/urine pregnancy test (WOCBP only) | X | X | X | X | X | X |
| Vital signs <sup>d</sup> | X | X | X | X | X | X |
| ECG | X | 40.000 | X | | | X |
| Targeted physical examination | X | X | X | X | X | X |
| Blood eosinophil count | X | | X | | X | X |
| Prebronchodilator FEV1 | X | | | | | |
| Postbronchodilator FEV1° | X | 4000 | | 10000 | | |
| Administration of benralizumab | | X | X | X | X | 200 |
| Recording Use of concomitant as thma<br>medication (OCS/ICS/LABA) | X | X | X | X | X | X |
| Adverse events and Serious adverse events <sup>f</sup><br>(reported <sup>g</sup> and observed) | Х | X | X | X | X | X |
| Assessment of asthma exacerbations | X | X | X | X | X | X |

Abbreviations: BMI = body mass index; EOS = end of study; ECG= Electrocardiogram; FEV1 = forced expiratory volume in one second; ICS = inhaled corticosteroid; LABA = long-acting beta-agonist; OCS = oral corticosteroid; UPT = urine pregnancy test; WOCBP = women of childbearing potential (after menarche)

- a. Recheck clinical status before first dose of benralizumab.
- b. Clinical safety laboratory assessment will include clinical chemistry, haematology, and urinalysis. Clinical chemistry will include serum alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, lactate dehydrogenase, total protein, total bilirubin, albumin, and serum creatinine. Haematology will include haematocrit, leucocyte count, leucocyte differential count (absolute count), platelet count, and haemoglobin. Urinalysis (dipstick) will assess urine haemoglobin/erythrocytes/blood, protein/albumin, and glucose.
- c. Serum pregnancy test will be done at baseline and UPT will be done at Day 1, Week 4, 8, 16, 24.
- d. The vital signs (pulse, blood pressure, respiration rate, and body temperature) will be taken before benralizumab administration, and, if possible, blood drawing and usual asthma controller medication. If it is



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

not logistically possible, sufficient time as per clinician discretion should be allotted between phlebotomy and vital signs assessment. For details, please refer to Section 8.1.3.

- e. When historical proof of postbronchodilator reversibility in FEV1 is not documented within 12 months before Visit 1, the reversibility test by spirometry will need to be performed either during screening or on Day 1 before first dose.
- f. While on study drug treatment and within 2 months after the end of study treatment/discontinuation of the study drug.
- g. Participants will be provided a patient diary to record any undesirable health-related experience or adverse events occurring during the study. Adverse events and serious adverse events mentioned both in the patient diary and verbally communicated by the participant will be recorded.

#### 2.3 Randomization

Not Applicable

### 2.4 Blinding and Un-Blinding

Not Applicable

#### 2.5 Interim Analysis

No interim analyses is planned for this study.

# 3. Population Analysis Set

#### 3.1 Enrolled Analysis Set

"Enrolled" means a participant's, or their legally authorised representative's, agreement by signing the ICF to participate in a clinical study following completion of the informed consent process.

#### 3.2 Assigned to Study intervention Analysis Set

Potential participants who fulfil the eligibility criteria and are assigned with the study identification number.

# 3.3 Evaluable Analysis Set

All participants assigned to study intervention and receiving at least 1 dose of study intervention and provide at least one post baseline assessment.

#### 3.4 Safety Analysis Set

All participants assigned to study intervention and who take at least 1 dose of study intervention.

#### 4. Sample Size and Power Calculations

The primary objective of this study is to assess safety and tolerability of benralizumab in adult (18 to 75 years of age) male or female patients who have severe asthma with eosinophilic phenotype requiring high dose of ICS and LABA.

| Document Pag |
|-------------------------------------------|
|-------------------------------------------|



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Based on the literature review, the below table is created for listing the key AEs (headache, pyrexia, pharyngitis and injection site reactions) and hypersensitivity reactions (e.g. anaphylaxis, angioedema, urticaria, urticaria papular, rash) which were included in the USPI, SmPC and the India PI, all in the range of 1% to 10%.

| | Incidence Rate (%) | | |
|--------------------------|--------------------|------|---------|
| Key AE Terms | SmPC/ India label | USPI | SIROCCO |
| Headache | | 8% | 7%-9% |
| Pharyngitis | 1 - | 5% | 4%-6% |
| Pyrexia | Common (1%-10%) | 3% | 3%-4% |
| Injection site reactions | | 2.2% | 2%-4% |
| Hypersensitivity | 1 - | 3% | 3% |

Effectiveness 
$$n = \frac{Z^2 P (1-P)}{d^2}$$

where n = calculated sample size, Z = tabulated Z statistic value for  $\alpha$  level of confidence, P = expected proportion of AEs and d = absolute precision level (half-width of the confidence interval [CI]).

Considering the maximum limit of the incidence rate of AEs to be 10%, approximately 139 evaluable participants will be required to present 95% CI around the estimated AE incidence rate with absolute precision level of 0.05. Considering dropout rate of 5%, a total of 147 participants will be required to be enrolled into the study.

# 5. Patient Characteristics and Study Conduct Summaries

#### 5.1 General Considerations

Statistical Analysis will be performed using SAS (version 9.4 or higher) software (SAS Institute Inc USA). Categorical variables will be summarized with the frequency, percentage of Patients in each category and corresponding 95% CI (using Clopper-Pearson exact Method, where appropriate). Continuous variables will be summarized descriptively with the number of Patients, mean, standard deviation, median, 25th and 75th percentiles and minimum and maximum values.

### 5.2 Decimal Point

Unless otherwise noted, means, median, will be presented to one decimal place more than the measured value, the same decimal as the measured value, percentages, 25th and 75th percentiles and 95% confidence intervals will be presented to two decimal places and p-value will be presented to three decimal place. Percentages after zero counts will not be displayed and percentages equating to 100% will be presented as 100%, without any decimal places.

### 5.3 Disposition of Patients

Patient disposition table will be based on all Evaluable Analysis Set who consented to participate in the study. The following summaries will be included in the disposition table: total number of Patient Enrolled in the study, total



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

number of Patients screened in the study, number of Patients who failed screening, number and percentage of Patients who completed the study and number and percentage of Patients who discontinued from the study with reason for discontinuation.

### 5.4 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized based on the Evaluable Analysis Set.

Descriptive summaries will be provided for the demographic and baseline characteristics. Demographic characteristics and baseline characteristics such as age, Gender and Race, etc. will be summarized and tabulated for Evaluable Analysis Set.

All the continuous variables will be summarized by n, mean, standard deviation, median, 25th and 75th percentiles and minimum and maximum values. All the categorical variables will be summarized as frequency, percentage of Patients in each category and corresponding 95% CI (using Clopper-Pearson exact Method, where appropriate).

#### 5.5 Covid-19 Vaccination

Covid-19 Vaccination will be summarized based on the Evaluable Population.

Descriptive summaries will be provided for the Covid-19 Vaccination.

All the continuous variables will be summarized by n, mean, standard deviation, median, 25th and 75th percentiles and minimum and maximum values. All the categorical variables will be summarized as frequency, percentage of Patients in each category and corresponding 95% CI (using Clopper-Pearson exact Method, where appropriate).

# 5.6 Medical History

Medical History will be summarized based on the Evaluable Population.

Descriptive summaries will be provided for the Medical History.

All the continuous variables will be summarized by n, mean, standard deviation, minimum, median and maximum values. All the categorical variables will be summarized as frequency, percentage of Patients in each category and corresponding 95% CI (using Clopper-Pearson exact Method, where appropriate).

#### 5.7 Electrocardiogram (ECG)

Electrocardiogram will include Heart rate, QRS, PR, RR, QT, QTcB. Electrocardiogram will be summarized based on the Safety Analysis Set.

Descriptive summaries will be provided for the Electrocardiogram.

All the continuous variables will be summarized by n, mean, standard deviation, median, 25th and 75th percentiles and minimum and maximum values. All the categorical variables will be summarized as frequency, percentage of Patients in each category and corresponding 95% CI (using Clopper-Pearson exact Method, where appropriate).



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# 6. Endpoints Analysis Strategy

# 6.1 Endpoints Analysis

# 6.1.1 Primary Endpoint

- Percentage of AEs, SAEs and TEAEs
- Nature, Incidence and Severity of AES, Including unexpected adverse drug reactions
- Percentage of patients with AEs that lead to Study treatment discontinuations or modifications

#### 6.1.2 Secondary Endpoint

- Time to first asthma exacerbation
- Annualised exacerbation rate
- Overall investigators assessment on the outcome of the treatment: "well controlled", "Partly Controlled" and
   "Uncortolled"
- Change in blood eosinophil levels from baseline at week 4, 16 and 24.

#### 6.2 Efficacy Hypothesis

There is no statistical hypothesis to be tested in this study.

# 6.3 Statstical Methods for Efficacy Analsysis

Statistical Analysis will be performed using SAS (version 9.4 or higher) software (SAS Institute Inc USA). Categorical variables will be summarized with the frequency and percentage of Patients in each category. Continuous variables will be summarized descriptively with the number of Patients, mean, standard deviation, 25th and 75th percentiles, minimum, median and maximum values.

### 6.3.1 Primary Endpoint Analysis

The primary analysis for primary endpoint will be based on Safety Analsysis Set.

Primary Endpoint evaluations will include Adverse Events (AEs), Serious Adverse Events (AEs), Treatment Emergent Adverse Event (TEAEs), Participants with unexpected Adverse Drug Reactions (ADRs) and Participants with AEs that lead to study treatment discontinuations or modifications.

Adverse Events (AEs), Serious Adverse Events (AEs), Treatment Emergent Adverse Event (TEAEs), Participants with unexpected Adverse Drug Reactions (ADRs) and Participants with AEs that lead to study treatment discontinuations or modifications will be summarized using Frequency, Percentages and 95% CIs (using Clopper-Pearson Exact method).



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

The AE profiles in participants will be presented as summaries showing the number of participants (n, %) along with number of events by System Organ Class and Preferred Terms assigned to the event by Medical Dictionary for Regulatory Activities (MedDRA) for the following:

- TEAEs
- SAEs
- Related and non-related TEAEs
- Serious and non-serious TEAEs
- TEAEs based on severity (Mild, Moderate, Severe)
- Unexpected ADRs based on severity (Mild, Moderate, Severe)

Physical Examination will include General Appearance, Respiratory system, Cardiovascular system, Abdomen, Skin, Head, Eye, Ear, Nose, Throat, Lymph node, Thyroid, Musculoskeletal system and Neurological System. Physical Examination will be summarized based on the Safety Analysis Set.

Descriptive summaries will be provided for the Physical Examination.

All the continuous variables will be summarized by n, mean, standard deviation, minimum, median and maximum values. All the categorical variables will be summarized as frequency, percentage of Patients in each category and corresponding 95% CI (using Clopper-Pearson exact Method, where appropriate).

Vital Signs will include Pulse rate, Respiratory rate, Systolic Blood Pressure, Diastolic Blood Pressure and Temperature.

Vital Signs will be summarized based on the Safety Analysis Set.

Vital Signs will be will be summarised descriptively for actual values and change from baseline values for each visit using the number of observations, arithmetic mean, SD, median, 25th and 75th percentiles, and minimum and maximum values.

The Vital signs (Pulse rate, Respiratory rate, Systolic Blood Pressure, Diastolic Blood Pressure and Temperature) in this study is to evaluate the change from baseline to Post-baseline will be analysed using Paired t – test / Wilcoxon signed-rank test at 5% level of significance.

Change from baseline will be determined as:

Change from Baseline = (Post-baseline - Baseline)

Percent Change Change from Baseline = ([Post-baseline - Baseline] / Baseline) X 100

Clinical Safety laboratory Assessment will include clinical chemistry, haematology and urinalysis. Clinical Safety laboratory assessment will be summarized based on the Safety Analysis Set.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Clinical Safety laboratory Assessment will be summarised descriptively for actual values and change from baseline values for each visit using the number of observations, arithmetic mean, SD, median, 25th and 75th percentiles, and minimum and maximum values.

The Clinical Safety Laboratory (If available) in this study is to evaluate the change from baseline to Post-baseline will be analysed using Paired t – test / Wilcoxon signed-rank test at 5% level of significance.

Change from baseline will be determined as:

Change from Baseline = (Post-baseline - Baseline)

Percent Change Change from Baseline = ([Post-baseline - Baseline] / Baseline) X 100

#### 6.3.2 Secondary Endpoint Analysis

All Secodary Endpoints will be summarized based on the Evaluable Analysis Set.

Descriptive summaries will be provided for the Asthma Exacerbation. All the continuous variables will be summarized by n, mean, standard deviation, minimum, median and maximum values. All the categorical variables will be summarized as frequency, percentage of Patients in each category and corresponding 95% CI (using Clopper-Pearson exact Method, where appropriate).

Time from first dose of study treatment to the first asthma exacerbation will be calculated as follows: Start Date of first asthma exacerbation minus Date of first dose of study treatment plus 1. The time to first asthma exacerbation for participants who do not experience an asthma exacerbation during the study period will be censored at 24 weeks, or at the time point after which an exacerbation could not be assessed (for lost-to-follow-up participants). The data will be summarised through median time to the first asthma exacerbation along with the 95% CI of median (as per availability of data) and displayed graphically using a KM plot.

Blood Eosinophils level will be summarized based on the Evaluable Analysis Set.

Blood Eosinophils will be summarised descriptively for actual values and change from baseline at week 4, 16, 24 using the number of observations, arithmetic mean, SD, median, 25th and 75th percentiles, and minimum and maximum values.

The Blood Eosinophils in this study is to evaluate the change from baseline to Post-baseline will be analysed using Paired t – test / Wilcoxon signed-rank test at 5% level of significance.

Change from baseline will be determined as:

Change from Baseline = (Post-baseline - Baseline)

Percent Change Change from Baseline = ([Post-baseline - Baseline] / Baseline) X 100

Overall Investigators Assessment will be summarized based on the Evaluable Analysis Set.

Descriptive summaries will be provided for the Overall Investigators Assessment.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

All the categorical variables will be summarized as frequency, percentage of Patients in each category and corresponding 95% CI (using Clopper-Pearson exact Method, where appropriate).

# 7. References

- 1. ICH E3 Guideline\_International Council for Harmonisation
- 2. ICH E9; STATISTICAL PRINCIPLES FOR CLINICAL TRIALS



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

### 8. Mock Tables

Table 14.1.1.1. Patient Disposition in the Study (Enrolled Analysis Set)

| | N = xx |
|-----------------------------------------|------------|
| | n (%) |
| Patients Enrolled/ Screened | XX |
| Evaluable Analysis Set | XX |
| Screen Failures | xx |
| Patients Completed the study | xx (xx.xx) |
| Patients Discontinued the study | xx (xx.xx) |
| Reason for Discontinuation/ Withdrawal | |
| Patient Decision | xx (xx.xx) |
| Adverse Event | xx (xx.xx) |
| Severe non-compliance to Study protocol | xx (xx.xx) |
| Disease Progression | xx (xx.xx) |
| Pregnancy or intent to become pregnant | xx (xx.xx) |
| Lost to Follow-up | xx (xx.xx) |
| Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other 2 | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Enrolled Analysis Set.
- The small "n" in summary statistics represents the total number of patients in the row category.
- Percentages in the "Patient completed the study" and "Patients Discontinued the study" rows are based on the total number of Enrolled Analysis Set.
- Percentages in the "Reasons for Discontinuation" rows are based on the number of Patients Discontinued study.
- There were 154 total enrolled/screened patients, 10 screen failures, 124 study completions, 20 trial discontinuations, however only 138 individuals were deemed eligible for analysis set because six patients meet the eligibility requirements but do not get the medication.
- Note: Screened Patients are those who signed the informed consent.
- Source: Listing 16.1.1.1 and Listing 16.1.1.3



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.1.2. Summary of Patient Discontinuation of Study Intervention (Evaluable Analysis Set )

| | N = xx<br>n (%) |
|---|---|
| Study Treatment stopped permanently before the scheduled treatment period | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Patient continuing in the study | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Reason for Withdrawal | |
| Patient Decision | xx (xx.xx) |
| Development of any study-specific criteria for discontinuation | xx (xx.xx) |
| Anaphylactic reaction to benralizumab requiring administration of epinephrine | xx (xx.xx) |
| Development of helminth parasitic infestations requiring hospitalisation | xx (xx.xx) |
| Intensive care unit admission with prolonged intubation and mechanical ventilation for asthma-related | |
| event | xx (xx.xx) |
| Severe non-compliance to study protocol | xx (xx.xx) |
| Eligibility criteria not met | xx (xx.xx) |
| Pregnancy or intent to become pregnant | xx (xx.xx) |
| Lost to follow-up | xx (xx.xx) |
| Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other 2 | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients in the row category.
- Percentages in the "Study treatment stopped permanently before the scheduled treatment period" rows are based on the total number of Evaluable Analysis Set.
- Percentages in the "Patient continuing in the study" and "Reason for Withdrawal" rows are based on the number of patients who stopped the study treatment permanently.
- Source: Listing 16.1.1.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.1.3. Summary of Analysis Population (Enrolled Analysis Set)

| | N = xx |
|------------------------|------------|
| | n (%) |
| Enrolled Analysis Set | xx (xx.xx) |
| Evaluable Analysis Set | xx (xx.xx) |
| Safety Analysis Set | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Enrolled Analysis Set.
- The small "n" in summary statistics represents the total number of patients in the row category.
- Percentages in the "Safety Population" row is based on the total number of Enrolled Analysis Set.
- Enrolled Analysis Set: "Enrolled" means a participant, or his/her legally authorised representative, agreed by signing the ICF to participate in a clinical study following completion of the informed consent process.
- Evaluable analysis Set: All participants assigned to study intervention and receiving at least 1 dose of study intervention and provide at least one post baseline assessment.
- Safety Population: All participants assigned to study intervention and who take at least 1 dose of study intervention.
- Source: Listing 16.1.1.4

Table 14.1.2.1. Summary of Demographic and Baseline Characteristics (Evaluable Analysis Set)

| Demographic and Baseline Variables | N = xx |
|--------------------------------------------------|----------------|
| Age (Years) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) |
| Gender | |
| Male | xx (xx.xx) |
| Female | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Female, Indicate childbearing potential | |
| Premenarchal | xx (xx.xx) |
| Premenopausal female | xx (xx.xx) |
| Postmenopausal female | xx (xx.xx) |
| Potentially able to bear children | xx (xx.xx) |
| Race | |
| Asian | xx (xx.xx) |
| Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other n | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- Percentages are based on number of Enrolled Analysis Set.
- SD = Standard Deviation, min=minimum, max=maximum
- Source: Listing 16.1.2.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.2.2. Summary of Anthropometric Assessment (Evaluable Analysis Set)

| | N = xx |
|--------------------------------------------------|----------------|
| Height (cm) | |
| n | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) |
| Weight (Kg) | |
| n | XX |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) |
| Body Mass Index (Kg/m²) | |
| n | XX |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- SD = Standard Deviation, min=minimum, max=maximum
- Source: Listing 16.1.2.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.3. Summary of Significant Medical History (Evaluable Analysis Set)

| System Organ Class /Preferred Term | N = xx |
|------------------------------------|------------|
| | n (%) |
| Patient with any medical history | xx (xx.xx) |
| System Organ Class 1 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |
| System Organ Class 2 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |
| System Organ Class 3 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |
| System Organ Class 4 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |
| System Organ Class 5 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients in the row category.
- All Percentages rows are based on number of Evaluable Analysis Set.
- Medical histories were coded using MedDRA Ver24.1
- Source: Listing 16.1.3



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.4. Summary of COVID-19 vaccination (Evaluable Analysis Set)

| | N = xx |
|---------------------------------------|------------|
| | n (%) |
| Patient received COVID-19 Vaccination | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| If Vaccination | |
| 1 <sup>st</sup> Dose | xx (xx.xx) |
| 2 <sup>nd</sup> Dose | xx (xx.xx) |
| 3 <sup>rd</sup> Dose | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients in the row category.
- Percentages in the "Patients received COVID-19 Vaccination" rows are based on the total number of Evaluable Analysis Set.
- Percentages in the "If Vaccination" rows are based on the total number of "Patient received covid-19 vaccination".
- Source: Listing 16.1.4



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.5.1. Summary of Prior Asthma Therapy (Evaluable Analysis Set)

| | N = xx |
|---|---|
| | n (%) |
| Patient take any prior asthma medication(s) other than oral/inhaled | Corticosteroid |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients in the row category.
- Percentages in the "Patient take any prior asthma medication(s) other than oral/inhaled Corticosteroid" rows are based on the total number of Evaluable Analysis Set.
- Source: Listing 16.1.5.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.5.2. Summary of oral/inhaled Corticosteroid (Evaluable Analysis Set)

| | N = xx |
|-------------------------------------------------------|------------|
| | n (%) |
| Patient receive any prior oral/inhaled Corticosteroid | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients in the row category.
- Percentages in the "Patient receive any prior oral/inhaled Corticosteroid" rows are based on the total number of Evaluable Analysis Set.

Source: Listing 16.1.5.2



| D | ocument Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|--------------|---------|
| | Effective Date: | 25-Nov-2021 | |

# Table 14.1.6. Patient Administration of Benralizumab (Evaluable Analysis Set)

| | N = xx |
|------------------------------------------------------------|------------|
| | n (%) |
| Visit x | |
| Patient administer study Medication at this visit (N*=xxx) | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients in the row category.
- All percentages are based on N\* i.e. the total number of patients of Evaluable Analysis set at the visit.
- Programmer Note: Visit x- Visit 1, Visit 2 and visit 3
- Source: Listing 16.1.6.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.7. Summary of Overdose (Evaluable Analysis Set)

| | N = xx |
|-----------------------------------------|------------|
| | n (%) |
| Overdose of study intervention recorded | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Adverse Event occurred due to overdose | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Overdose Accidental | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients in the row category.
- All percentages are based on the Evaluable Analysis set.
- Source: Listing 16.1.6.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.8. Summary of Pulmonary Function Test (Evaluable Analysis Set)

| | N = xx |
|---|---|
| Pulmonary function test using Spirometer performed | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Pre-Bronchodilator Assessment | |
| Forced Expiratory Volume in 1 second (L) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) |
| redicted Normal FEV1 (%) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) |
| Forced Vital Capacity (L) | (canal, canal, |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) |
| Patient have historical proof of Post-Bronchodilator reversibility within 12 months | (^^.^^, ^^.^^) |
| Yes | vv (vv vv) |
| | xx (xx.xx) |
| No<br>Mississ | xx (xx.xx) |
| Missing | xx (xx.xx) |
| orced expiratory volume in 1 Second (L) | V |
| n<br>Maria | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) |
| Reversibility FEV1 (%) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) |
| FEV1 Reversibility (mL) | |
| n | Xx |
| Document | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Missing | Xx |
|--------------------------------------------------|----------------|
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- Percentages are based on number of Evaluable Analysis Set.
- SD = Standard Deviation, min=minimum, max=maximum
- Source: Listing 16.1.7



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.1.1. Summary of Asthma and Exacerbation (Evaluable Analysis Set)

| | N = xx<br>n (%) | 95% CI |
|---|---|---|
| Visit 1 | | |
| Significant History of Asthma with Eosinophilic Phenotype | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| Missing | xx (xx.xx) | (xx.xx, xx.xx) |
| Disease Duration (months) | | |
| n | Xx | |
| Missing | Xx | |
| Mean (SD) | xx.x (xx.xx) | |
| Median | xx.x | |
| (min, max) | (xx.xx, xx.xx) | |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) | |
| Patient Experience Exacerbation in the previous 12 months | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| Missing | xx (xx.xx) | (xx.xx, xx.xx) |
| Visit x | | |
| Patient Experience any new Exacerbation or change in existing Exacerbation since last visit | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| Missing | xx (xx.xx) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- All Percentages rows are based on the total number of Evaluable Analysis Set.
- 95% CI calculate will be using Clopper-Pearson Exact method.
- Programmer Note: Visit x- Visit 2, Visit 3, Visit 4 and Visit 5
- Source: Listing 16.2.1.1 and Listing 16.2.1.2


| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.1.2. Summary of Exacerbation (Evaluable Analysis Set)

| | N = xx | |
|---|---|---|
| | n (%) | 95% CI |
| Outcome | | |
| Resolved | xx (xx.xx) | (xx.xx, xx.xx) |
| Fatal | xx (xx.xx) | (xx.xx, xx.xx) |
| Not Resolved | xx (xx.xx) | (xx.xx, xx.xx) |
| Patient withdrawn due to exacerbation | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| Exacerbation is Clinical Significance | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| Patient visit the Emergency room due to this Exacerbation | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| If Yes, Number of Telephone calls | | |
| n | Xx | |
| Missing | Xx | |
| Mean (SD) | xx.x (xx.xx) | |
| Median | xx.x | |
| (min, max) | (xx.xx, xx.xx) | |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) | |
| Patient Hospitalisation due to this Exacerbation | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| Patient visit to clinic as out-patient | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| Oral/Inhaled Corticosteroids taken for the Exacerbation | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| Patient intubated for this exacerbation | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| Exacerbation medications other than oral/inhaled | | |
| Corticosteroids taken | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of Events.
- Percentages are based on the number of Evaluable Analysis Set
- 95% CI calculate will be using Clopper-Pearson Exact method.
- \*Patient 09021 is counted under both 'Yes' and 'No'. The patient had 4 exacerbation events. It had visited the emergency room for 1 exacerbation event but not visited the emergency room for other 3 events.
- Source: Listing 16.2.2.1, Listing 16.2.2.2 and Listing 16.2.2.3



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.1.3. Summary of Before and After Treatment Exacerbation (Evaluable Analysis Set)

| | N = xx |
|---------------------------------------|--------------|
| Exacerbation | |
| before study | |
| N | XX |
| Missing | XX |
| Mean (SD) | x.x (x.xx) |
| Median | x.x |
| (min, max) | (x,x) |
| (25th Percentile,<br>75th Percentile) | (x.xx, x.xx) |
| Exacerbation at<br>end of study | |
| n | xx |
| Missing | xx |
| Mean (SD) | x.x (x.xx) |
| Median | x.x |
| (min, max) | (x,x) |
| (25th Percentile,<br>75th Percentile) | (x.xx, x.xx) |
| P-value | x.xxxx |
| Annualized<br>exacerbation | x.xx |
| rate | |

- The column header's capital "N" denotes the total number of Evaluable Analysis Sets.
- The modest "n" in the number of patients suffering from exacerbation.
- The annual rate for each patient was calculated by dividing the total number of exacerbations by the number of days participated in the study and multiplying by 365.
- Source: Listing 16.2.2.1, Listing 16.2.2.2 and Listing 16.2.2.3



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.2. Summary of Time to first Exacerbation (Evaluable Analysis Set)

| | N=xxx |
|------------------------------------------------------------|----------------|
| Patient Asthma Exacerbation, n (%) | |
| Yes | xx(xx.xx) |
| No | xx(xx.xx) |
| Duration of Patient First Asthma Exacerbation (Days) | |
| n | Xx |
| missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min , max ) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> Percentile, 75 <sup>th</sup> Percentile) | (xx.xx, xx.xx) |
| Estimate for Time to Response (Days) | |
| Median | xx.x |
| 95 % CI | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients
- Estimate for Time to Response using Kaplan-Meier method.
- Start date of first asthma exacerbation minus Date of First dose of study treatment Plus 1.
- Source: Listing 16.2.2.1, Listing 16.2.2.2 and Listing 16.2.2.3



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.3. Analysis of change in Blood Eosinophils count from baseline to Visit 2, Visit 4 and Visit 5 (Evaluable Analysis Set)

| | Observed value | Change from Baseline | % Change from Baseline |
|---|---|---|---|
| | (N = xx) | (N = xx) | (N = xx) |
| Absolute Eosinophil | | | |
| Baseline (Screening Visit) | | | |
| n | XX | | |
| Missing | xx | | |
| Mean (SD) | xx.x (xx.xx) | | |
| Median | xx.x | | |
| (min, max) | (xx.xx, xx.xx) | | |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) | | |
| Visit x | | | |
| n | XX | XX | XX |
| Missing | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75th percentiles) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| p-value | | x.xxx | x.xxx |

- The Capital "N" in the column header represents the total number of Patients in Safety Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- SD = Standard deviation, min=minimum, max=maximum
- Change from Baseline Post-Baseline Baseline
- % Change from Baseline = (Post-Baseline Baseline / Baseline) X 100
- p-value calculate using paired t test.
- Programmer Note: Visit x: Visit 2, Visit 4 and Visit 5
- Source: Listing 16.2.3



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.4 Summary of Overall Investigators Assessment (Evaluable Analysis Set)

| | N = xx | |
|--------------------------------------------|------------|----------------|
| | n (%) | 95% CI |
| Overall Investigators Assessment performed | | |
| Yes | xx (xx.xx) | (xx.xx, xx.xx) |
| No | xx (xx.xx) | (xx.xx, xx.xx) |
| If yes | | |
| Well Controlled | xx (xx.xx) | (xx.xx, xx.xx) |
| Partly Controlled | xx (xx.xx) | (xx.xx, xx.xx) |
| Uncotrolled | xx (xx.xx) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of Evaluable Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- Percentages in the "Overall Investigators Assessment performed" rows are based on the total number of Evaluable Analysis Set.
- Percentages in the "If Yes" rows are based on the total number of "Patient Performed overall Investigation Assessment".
- 95% CI calculate will be using Clopper-Pearson Exact method.
- Source: Listing 16.2.4



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.1.1. Overall Summary of Adverse Events (Safety Analysis Set)

| | (N=xx) |
|---------------------------------------------------|---------------|
| | n (%) E |
| Patient with at least one AE | xx (xx.xx) xx |
| Patients with at least one Serious AE | xx (xx.xx) xx |
| Patient with at least one TEAE | xx (xx.xx) xx |
| Patients with at least one Serious TEAE | xx (xx.xx) xx |
| Subjects with at least drug related TEAE | xx (xx.xx) xx |
| Patients with any TEAE Leading to discontinuation | xx (xx.xx) xx |
| Patients with any TEAE Leading to death | xx (xx.xx) xx |

- TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set
- n = number of patients in row category.
- TEAE are those adverse events which occurred after first dose of study medication.
- All Percentage rows are based on the Safety Analysis Set.
- Note: Adverse events were coded using MedDRA version 24.1 If a Patient has multiple occurrences of an AE, the Patient is
  presented only once in the respective patient count column (n) for the corresponding AE. Events are counted each time in
  the event (E) column.
- Source: Listing 16.3.1.2, Listing 16.3.2.1 and Listing 16.3.2.2



| Document Title: | Document ID: | BP04-01 |
|----------------------------|-----------------|-------------|
| Chattataal Assalasta Blass | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.3.1.2. Summary of Treatment Emergent Adverse Events (Safety Analysis Set)

| | (N=xx) | |
|---|---|---|
| | n (%) E | 95% CI |
| Adverse Events | | |
| Patient with any TEAE | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Patient with any Serious TEAE | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Adverse Events by Intensity grade | | |
| Mild | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Moderate | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Severe | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Action Taken | | |
| None | xx (xx.xx) xx | (xx.xx, xx.xx) |
| None-drug treatment required | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Hostpitalisation/prolonged hostpitalisation | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Diagnostic or clinical test conducted | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Drug withdrawn | xx (xx.xx) xx | (xx.xx, xx.xx) |
| TEAE by outcome | | |
| Recovered without sequelae | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Recovered with Sequelae | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Not recovered/Not resolved | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Recovering/Resolving | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Unknown | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Fatal | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Investigators causality rating against the Investigational Product | | |
| Yes | xx (xx.xx) xx | (xx.xx, xx.xx) |
| No | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Patient Withdrawn | | |
| Yes | xx (xx.xx) xx | (xx.xx, xx.xx) |
| No | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Non-Study Medication Teatment taken | , , | |
| Yes | xx (xx.xx) xx | (xx.xx, xx.xx) |
| No | xx (xx.xx) xx | (xx.xx, xx.xx) |

- TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis
- n = number of patients in row category, E = number of TEAE.
- TEAE are those adverse events which occurred after first dose of study medication.
- All Percentages rows are based on the total number of patients in the Safety Analysis Set
- 95% CI calculate will be using Clopper-Pearson Exact method.
- Source: Listing 16.3.1.2



| Document Title: | Document ID: | BP04-01 |
|----------------------------|-----------------|-------------|
| Chattataal Assalasta Blass | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.3.1.3.1 Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set)

| | (N=xx) |
|-----------------------------------|---------------|
| System Organ Class/Preferred Term | n (%) E |
| Patient with at least one TEAE | xx (xx.xx) xx |
| System Organ Class | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |
| System Organ Class | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |

- TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set
- n = number of patients in row category; E = number of TEAE
- TEAE are those adverse events which occurred after first dose of study medication.
- All Percentages ros are based on the total number of patients in the Safety Analysis Set .
- System Organ classes was sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.
- Adverse events were coded using MedDRA version 24.1 If a patient has multiple occurrences of an AE, the
  patient is presented only once in the respective patient count column (n) for the corresponding AE. Events are
  counted each time in the event column.
- Source: Listing 16.3.1.2, Listing 16.3.2.1 and Listing 16.3.2.2



| Document Title: | Document ID: | BP04-01 |
|----------------------------|-----------------|-------------|
| Chattataal Assalasta Blass | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.3.1.3.2 Summary of Serious Treatment Emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set)

| | (N=xx) |
|----------------------------------------|---------------|
| System Organ Class/Preferred Term | n (%) E |
| Patient with at least one Serious TEAE | xx (xx.xx) xx |
| System Organ Class | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |
| System Organ Class | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |

- TEAE = treatment-emergent adverse event; N = number of Patients in the Safety Analysis Set
- n = number of patients in row category; E = number of TEAE
- TEAE are those adverse events which occurred after first dose of study medication.
- All Percentages ros are based on the total number of patients in the Safety Analysis Set .
- System Organ classes was sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.
- Adverse events were coded using MedDRA version 24.1 If a patient has multiple occurrences of an AE, the
  patient is presented only once in the respective patient count column (n) for the corresponding AE. Events are
  counted each time in the event column.
- Source: Listing 16.3.1.2, Listing 16.3.2.1 and Listing 16.3.2.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Dlaw | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.3.1.4. Summary of TEAE related to the Investigational Product by System Organ Class and Preferred Term (Safety Analysis Set)

| | (N=xx) |
|-----------------------------------------|---------------|
| System Organ Class/Preferred Term | n (%) E |
| Patient with any TEAE related to the IP | xx (xx.xx) xx |
| System Organ Class | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |
| System Organ Class | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |

- TEAE = treatment-emergent adverse event; N = number of patients in Safety Analysis Set
- n = number of Patients in row category; E = number of TEAE
- IP=Investigational product
- TEAE are those adverse events which occurred after first dose of study medication.
- All Percentage rows are based on the total number of patients in the Safety Analysis Set.
- System organ classes are sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class. Related includes possible and probable
- Adverse events were coded using MedDRA version 24.1. If a patient has multiple occurrences of an AE, the patient is
  presented only once in the respective patient count column (n) for the corresponding AE. Events are counted each time in
  the event € column.
- Source: Listing 16.3.1.2, Listing 16.3.2.1 and Listing 16.3.2.2



| Document Title: | Document ID: | BP04-01 |
|----------------------------|-----------------|-------------|
| Chattataal Assalasta Blass | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.3.1.5. Summary of TEAE leading to discontinuation by System Organ Class and Preferred Term (Safety Analysis Set)

| | (N=xx) | |
|---|---|---|
| System Organ Class/Preferred Term | n (%) E | 95% CI |
| Patient with any TEAE leading to discontinuation | xx (xx.xx) xx | (xx.xx, xx.xx) |
| System Organ Class | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Preferred Term 1 | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Preferred Term 2 | xx (xx.xx) xx | (xx.xx, xx.xx) |
| System Organ Class | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Preferred Term 1 | xx (xx.xx) xx | (xx.xx, xx.xx) |
| Preferred Term 2 | xx (xx.xx) xx | (xx.xx, xx.xx) |

- TEAE = treatment-emergent adverse event; N = number of patients in Safety Analysis Set; n = number of patients in row category; E = number of TEAE
- IP Investigartional product
- TEAE are those adverse events which occurred after first dose of study medication.
- All Percentages roes are based on the total number of patients in the Safety Analysis Set.
- System organ classes are sorted by descending frequency. Preferred terms are sorted by descending frequency overall
  within system organ class.
- Adverse events will be using MedRA version 24.1. If a patient has multiple occurrences of an AE, the patient is presented
  only once in the respective patient count column (n) for the corresponding AE. Events are counted each time in the event
  E column.
- 95% CI calculate will be using Clopper-Pearson Exact method.
- Source: Listing 16.1.4, Listing 16.3.1.2, Listing 16.3.2.1 and Listing 16.3.2.2



| Document Title: | Document ID: | BP04-01 |
|----------------------------|-----------------|-------------|
| Chattataal Assalasta Blass | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.3.1.6. Summary of Serious TEAE by System Organ Class and Preferred Term (Safety Analysis Set)

| | (N=xx) |
|----------------------------------------|---------------|
| System Organ Class/Preferred Term | n (%) E |
| Patient with at least one serious TEAE | xx (xx.xx) xx |
| System Organ Class | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |
| System Organ Class | xx (xx.xx) xx |
| Preferred Term 1 | xx (xx.xx) xx |
| Preferred Term 2 | xx (xx.xx) xx |

- TEAE = treatment-emergent adverse event; N = number of patients in Safety Analysis Set;
- n = number of Patients in row category; E = number of serious TEAE
- TEAE are those adverse events which occurred after first dose of study medication.
- All Percentages rows are based on the total number of patients in the Safety Analysis Set.
- System Organ classes was sorted by descending frequency. Preferred terms are sorted by descending frequency within system organ class.
- Adverse events were coded using MedDRA version 24.1 If a patient has multiple occurrences of an AE, the patient is
  presented only once in the respective patient count column (n) for the corresponding AE. Events are counted each time in
  the event € column.
- Source: Listing 16.3.1.2, Listing 16.3.2.1 and Listing 16.3.2.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.2.1. Analysis of change in Haematology parameters from baseline to Week 24. (Safety Analysis Set)

| | Observed value | Change from Baseline | % Change from Baseline |
|---|---|---|---|
| | (N = xx) | (N = xx) | (N = xx) |
| Haematology parameter x | | | |
| Baseline (Screening Visit) | | | |
| n | XX | | |
| Missing | xx | | |
| Mean (SD) | xx.x (xx.xx) | | |
| Median | xx.x | | |
| (min, max) | (xx.xx, xx.xx) | | |
| (25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | (xx.xx, xx.xx) | | |
| Week 24 | | | |
| n | XX | XX | XX |
| Missing | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| p-value | | x.xxx | x.xxx |

- The Capital "N" in the column header represents the total number of patients in Safety Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- SD = Standard deviation, min=minimum, max=maximum
- Change from Baseline Post-Baseline Baseline
- % Change from Baseline = (Post-Baseline Baseline / Baseline) X 100
- p-value calculate using paired t test.
- Programmer Note: Haematology parameter x: Haematocrit (%), Haemoglobin(g/DL), Absolute Neutrophils (mm³), Absolute Basophils(mm³), Absolute Eosinophils(mm³), Absolute Monocytes(mm³), Absolute Lymphocytes(mm³), Platelet count (/μL) and Total leukocyte count(/μL)
- Source: Listing 16.3.3.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.2.2. Analysis of change in Biochemistry parameters from baseline to Week 24 (Safety Analysis Set)

| | Observed value | Change from Baseline | % Change from Baseline |
|---|---|---|---|
| | (N = xx) | (N = xx) | (N = xx) |
| Biochemistry parameter x | | | |
| Baseline (Screening Visit) | | | |
| n | XX | | |
| Missing | xx | | |
| Mean (SD) | xx.x (xx.xx) | | |
| Median | xx.x | | |
| (min, max) | (xx.xx, xx.xx) | | |
| (25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | (xx.xx, xx.xx) | | |
| Week 24 | | | |
| n | Xx | Xx | xx |
| Missing | Xx | Xx | Xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| p-value | | x.xxx | x.xxx |

- The Capital "N" in the column header represents the total number of patients in Safety Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- SD = Standard deviation, min=minimum, max=maximum
- Change from Baseline Post-Baseline Baseline
- % Change from Baseline = (Post-Baseline Baseline / Baseline) X 100
- p-value calculate using paired t test.
- Programmer Note: Biochemistry parameter x: Serum Alkaline phosphatase (IU/L), Alanine aminotransferase(U/L), Aspartate aminotransferase (U/L), Gamma- glutamyl transferase(U/L), Lactate dehydrogenase(U/L), Total Protein (g/dL), Total bilirubin (mg/dL), Albumin (g/dL), Serum Creatinine (mg/dL).
- Source: Listing 16.3.3.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.3. Analysis of change in Vital Sign parameters from baseline to Visit 1, Visit 2, Visit 3, Visit 4 and Visit 5 (Safety Analysis Set)

| | Observed value | Change from Baseline | % Change from Baseline |
|---|---|---|---|
| | (N = xx) | (N = xx) | (N = xx) |
| Vital Sign parameter x | | | |
| Baseline (Screening Visit) | | | |
| n | XX | | |
| Missing | xx | | |
| Mean (SD) | xx.x (xx.xx) | | |
| Median | XX.X | | |
| (min, max) | (xx.xx, xx.xx) | | |
| (25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | (xx.xx, xx.xx) | | |
| Visit x | | | |
| n | Xx | Xx | xx |
| Missing | Xx | Xx | Xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| p-value | | x.xxx | x.xxx |

- The Capital "N" in the column header represents the total number of patients in Safety Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- SD = Standard deviation, min=minimum, max=maximum
- Change from Baseline Post-Baseline Baseline
- % Change from Baseline = (Post-Baseline Baseline / Baseline) X 100
- p-value calculate using paired t test.
- Programmer Note: Vital Signs parameter x: Pulse rate (beats/min), Respiratory rate (breaths/min), Systolic blood pressure (mmHg), Diastolic blood pressure (mmHg) and Temperature(°F).
- Programmer Note: Visit x: Visit 1, Visit 2, Visit 3, Visit 4 and Visit 5
- Source: Listing 16.3.4



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Version Number: | 3.1 | |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.3.4. Summary of Electrocardiogram (Safety Analysis Set)

| | N = xx |
|---|---|
| Visit x | |
| ECG performed | and the send |
| Yes<br>No | xx (xx.xx) |
| Heart Rate (beats/min) | xx (xx.xx) |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | (xx.xx, xx.xx) |
| QRS (ms) | (^^,^, ^^, |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | (xx.xx, xx.xx)<br>(xx.xx, xx.xx) |
| PR (ms) | (^^.^^, ^^.^^) |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | (xx.xx, xx.xx) |
| RR (ms) | (^^,^, ^^, |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| (25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | |
| QT (ms) | (xx.xx, xx.xx) |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median Median | XX.X |
| (min, max)<br>(25 <sup>th</sup> percentiles, 75 <sup>th</sup> percentiles) | (xx.xx, xx.xx)<br>(xx.xx, xx.xx) |
| | (xx.xx, xx.xx) |
| QTcB (ms) | V. |
| N Missing | Xx |
| Missing Mean (SD) | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| Document | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

#### (25th percentiles, 75th percentiles)

(xx.xx, xx.xx)

- The Capital "N" in the column header represents the total number of patients in Safety Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- Percentages are based on number of Safety Analysis Set.
- SD = Standard Deviation, min=minimum, max=maximum
- Programmer Note: Visit x: Screening Visit, Visit 2 and Visit 5
- Source: Listing 16.3.5



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.5. Summary of Targeted Physical Examination (Safety Analysis Set)

| | N = xx |
|--------------------------------------|--------------|
| | n (%) |
| Visit x | |
| Physical Examination Performed | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| General Appearance | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Respiratory System | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Cardiovascular System | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Abdomen | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Skin | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | , , |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Head, Eye, Ear, Nose, Throat | , , |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | , , |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Lymph Node | ,, |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | (, |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Thyroid | iii (valial) |
| Normal | xx (xx.xx) |
| roprietary and Confidential Document | Page 54 o |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Abnormal | xx (xx.xx) |
|------------------------|------------|
| If Abnormal | , , |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Musculoskeletal System | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Neurological System | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Other | |
| Normal | xx (xx.xx) |
| Abnormal | xx (xx.xx) |
| If Abnormal | |
| Abnormal CS | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of patients in Safety Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- All Percentages rows are based on the total number of Safety Analysis Set.
- Programmer note: Visit x: Screening Visit, Visit 1, Visit 2, Visit 3, Visit 4 and Visit 5.
- Source: Listing 16.3.6



| D | ocument Title: | Document ID: | BP04-01 |
|----------------------------|-----------------|-----------------|---------|
| Statistical Applicate Disc | | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 | |

Table 14.3.6.1. Summary of Serum Pregnancy Test (Safety Analysis Set)

| | N = xx |
|--------------------------------|------------|
| | n (%) |
| Serum Pregnancy test performed | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Result | |
| Positive | xx (xx.xx) |
| Negative | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- All Percentages rows are based on the total number of Safety Analysis Set.
- Source: Listing 16.3.3.4



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.6.2. Summary of Urine Pregnancy Test (Safety Analysis Set)

| | N = xx |
|--------------------------------|------------|
| | n (%) |
| Visit x | |
| Urine Pregnancy test performed | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Result | |
| Positive | xx (xx.xx) |
| Negative | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Analysis Set.
- The small "n" in summary statistics represents the total number of patients.
- All Percentages rows are based on the total number of Safety Analysis Set.
- Programmer note: Visit x- Visit 1, Visit 2, Visit 3, Visit 4 and Visit 5
- Source: Listing 16.3.7



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Pla | Effective Date: | 25-Nov-2021 |

Listing 16.1.1.1. Listing of Patient Informed consent

| Patient No | Informed Consent Obtained | Date of Informed Consent obtained | Time of Informed Consent obtained |
|---|---|---|---|
| XX-XXX | Yes/No | DD-MMM-YYYY | HH:MM |
| XX-XXX | Yes/No | DD-MMM-YYYY | HH:MM |
| XX-XXX | Yes/No | DD-MMM-YYYY | HH:MM |
| XX-XXX | Yes/No | DD-MMM-YYYY | HH:MM |
| xx-xxx | Yes/No | DD-MMM-YYYY | HH:MM |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Pla | Effective Date: | 25-Nov-2021 |

# Listing 16.1.1.2. Listing of Patient Discontinuation of Study Intervention

| Patient | Study Treatment stopped permanently before | Patient Continue in | | Primary reason | If Other, |
|---|---|---|---|---|---|
| No | the scheduled end of treatment period | the Study | Date of Last Dose | for withdrawal | Specify |
| xx-xxx | Yes/No | Yes/No | DD-MMM-YYYY | Xxxx | Xxxx |
| XX-XXX | Yes/No | Yes/No | DD-MMM-YYYY | Xxxx | Xxxx |
| XX-XXX | Yes/No | Yes/No | DD-MMM-YYYY | Xxxx | Xxxx |
| xx-xxx | Yes/No | Yes/No | DD-MMM-YYYY | Xxxx | Xxxx |
| XX-XXX | Yes/No | Yes/No | DD-MMM-YYYY | XXXX | xxxx |



| | Document Title: | Document ID: | BP04-01 |
|-----------------------------|-----------------|-----------------|---------|
| Chabintinal Applicate Plans | | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 | |

# Listing 16.1.1.3. Listing of Patient Study Completion

| Patient | Patient complete | Patient complete Date of Completion/ Primary reason | | If Other, |
|---|---|---|---|---|
| No | the study | Discontinuation | withdrawal | Specify |
| XX-XXX | Yes/No | DD-MMM-YYYY | Xxxx | Xxxx |
| XX-XXX | Yes/No | DD-MMM-YYYY | Xxxx | Xxxx |
| XX-XXX | Yes/No | DD-MMM-YYYY | Xxxx | Xxxx |
| XX-XXX | Yes/No | DD-MMM-YYYY | Xxxx | Xxxx |
| XX-XXX | Yes/No | DD-MMM-YYYY | xxxx | xxxx |



| Document Title: | Document ID: | BP04-01 |
|-----------------|-----------------|---------|
| Effective Date: | 25-Nov-2021 | |

## Listing 16.1.1.4. Listing of Patient Analysis Set

| Patient | Enrolled Analysis | Assigned to study intervention | | |
|---|---|---|---|---|
| No | Set | Analysis Set | <b>Evaluable Analysis Set</b> | Safety Analysis Set |
| XX-XXX | Yes/No | Yes/No | Yes/No | Yes/No |
| xx-xxx | Yes/No | Yes/No | Yes/No | Yes/No |
| xx-xxx | Yes/No | Yes/No | Yes/No | Yes/No |
| XX-XXX | Yes/No | Yes/No | Yes/No | Yes/No |
| XX-XXX | Yes/No | Yes/No | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

### Listing 16.1.2.1. Listing of Patient Demographics Information

| Patient No | Date of Birth | Age (Years) | Gender | Indicate child-bearing potential | Date of last menses | Race | Other Specify |
|---|---|---|---|---|---|---|---|
| XX-XXX | DD-MMM-YYYY | Xx | Male/Female | xxxx | DD-MMM-YYYY | Asian/Other | XXXX |
| XX-XXX | DD-MMM-YYYY | XX | Male/Female | xxxx | DD-MMM-YYYY | Asian/Other | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Dlan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.1.2.2. Listing of Patient Anthropometry

| Patient No | Height (cm) | Weight (Kg) | Body Mass Index (Kg/m²) |
|------------|-------------|-------------|-------------------------|
| XX-XXX | XXX | XXX | xxx |
| XX-XXX | XXX | XXX | XXX |
| XX-XXX | XXX | XXX | XXX |
| XX-XXX | XXX | XXX | XXX |
| XX-XXX | XXX | XXX | xxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Applysis Plan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.1.3. Listing of Patient Significant Medical History

| | Patient have any | Seq. | Medical/Surgical | | | | Received |
|---|---|---|---|---|---|---|---|
| Patient No | medical/surgical History | No. | Description | Start Date | End Date | Ongoing | Treatment |
| XX-XXX | Yes/No | Xx | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | Yes/No |
| xx-xxx | Yes/No | XX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.1.4. Listing of Patient COVID-19 Vaccination

| Patient No | Patient received COVID-19 vaccine | Date of 1st Dose | Date of 2 <sup>nd</sup> Dose | Date of 3 <sup>rd</sup> Dose |
|---|---|---|---|---|
| XX-XXX | Yes/No | DD-MMM-YYYY/NA | DD-MMM-YYYY/NA | DD-MMM-YYYY/NA |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Applysis Plan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.1.5.1. Listing of Patient Prior Asthma Therapy

| Patient | Patient take any prior asthma medication | Seq. | Drug | | | | Total Daily | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| No | other than oral/Inhaled Corticosteroid | No. | name | Start Date | Stop Date | Ongoing | Dose | Units | Frequency | Route |
| XX-XXX | Yes/No | Xx | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | xxxx | XXXX | XXXX | XXXX |
| XX-XXX | Yes/No | XX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | xxxx | XXXX | xxxx | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

### Listing 16.1.5.2. Listing of Patient Prior Oral/Inhaled Corticosteroid Therapy

| Patient | Patient receive any oral/Inhaled | Seq. | Drug | | | | Duration | Total Daily | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| No | Corticosteroid therapy | No. | name | Start Date | Stop Date | Ongoing | (Years: Months) | Dose | Units | Frequency | Route |
| XX-XXX | Yes/No | XX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | xx : xx | xxxx | XXXX | XXXX | XXXX |
| XX-XXX | Yes/No | XX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | xx : xx | XXXX | XXXX | XXXX | XXXX |
| XX-XXX | Yes/No | XX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | xx : xx | XXXX | XXXX | XXXX | XXXX |
| XX-XXX | Yes/No | XX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | xx : xx | xxxx | XXXX | XXXX | XXXX |
| XX-XXX | Yes/No | XX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | xx : xx | xxxx | XXXX | XXXX | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.1.6.1. Listing of Patient Administration of Benralizumab

| Patient administer Study | | | | Date and time of Medication |
|---|---|---|---|---|
| Patient No | Visit | Medication at this visit | Dose | Administration |
| xx-xxx | Xxxx | Yes/No | 30 mg/mL | DD-MMM-YYYY/HH:MM |
| xx-xxx | Xxxx | Yes/No | 30 mg/mL | DD-MMM-YYYY/HH:MM |
| XX-XXX | Xxxx | Yes/No | 30 mg/mL | DD-MMM-YYYY/HH:MM |
| xx-xxx | Xxxx | Yes/No | 30 mg/mL | DD-MMM-YYYY/HH:MM |
| xx-xxx | Xxxx | Yes/No | 30 mg/mL | DD-MMM-YYYY/HH:MM |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

### Listing 16.1.6.2. Listing of Patient Overdose

| | Any Overdose of study | Any Adverse Event Occurred | Seq. | | Visit of | Overdose | Possible |
|---|---|---|---|---|---|---|---|
| Patient No | interventional recorded | due to Overdose | of AE | Date of Overdose | Overdose | Accidental | Cause |
| XX-XXX | Yes/No | Yes/No | Xx | DD-MMM-YYYY | Xx | Yes/No | Xxxx |
| XX-XXX | Yes/No | Yes/No | XX | DD-MMM-YYYY | xx | Yes/No | Xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.1.7. Listing of Patient Pulmonary Function Test

| | Pulmonary function | | | | | Patient have any historical | | Post- | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Patient | test using Spirometer | Date and Time of | Pre-Bronchodilator | | | proof of Post- Bronchodilator | Date of | Bronchodilator | | |
| No | performed | Assessment | of Assessment | Unit | Result | reversibility within 12 months | Assessment | of Assessment | Unit | Result |
| XX-XXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | Xxxx | Xxxx | Yes/No | Xxxx | Xxxx | Xxxx | Xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Flan | Effective Date: | 25-Nov-2021 |

Listing 16.2.1.1. Listing of Patient Asthma and Exacerbation History

| | Significant history of Asthma | | Disease Duration (Years: | Patient Experience exacerbation in the |
|---|---|---|---|---|
| Patient No | with Eosinophilic | Date of Diagnosis | Months) | previous 12 months |
| XX-XXX | Yes/No | DD-MMM-YYYY | YY:MM | Yes/No |
| XX-XXX | Yes/No | DD-MMM-YYYY | YY:MM | Yes/No |
| XX-XXX | Yes/No | DD-MMM-YYYY | YY:MM | Yes/No |
| xx-xxx | Yes/No | DD-MMM-YYYY | YY:MM | Yes/No |
| XX-XXX | Yes/No | DD-MMM-YYYY | YY:MM | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | | 25-Nov-2021 |

Listing 16.2.1.2. Listing of Patient Assessment of Asthma and Exacerbation

| | | Patient Experience any new exacerbation or change in |
|------------|-------|------------------------------------------------------|
| Patient No | Visit | exacerbation since last visit |
| xx-xxx | XXXX | Yes/No |
| xx-xxx | XXXX | Yes/No |
| xx-xxx | XXXX | Yes/No |
| xx-xxx | xxxx | Yes/No |
| xx-xxx | xxxx | Yes/No |


| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# Listing 16.2.2.1. Listing of Patient Exacerbation (Part 1)

| Patient | Seq. | | | Date of | | Primary Cause of | Patient withdrawn due to this | Exacerbation Clinical |
|---|---|---|---|---|---|---|---|---|
| No | No | Date of Onset | Outcome | Resolution | Date of Death | Exacerbation | Exacerbation | Significant |
| xx-xxx | Xx | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Xxxx | Yes/No | Yes/No |
| XX-XXX | Xx | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Xxxx | Yes/No | Yes/No |
| XX-XXX | Xx | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Xxxx | Yes/No | Yes/No |
| xx-xxx | Xx | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Xxxx | Yes/No | Yes/No |
| xx-xxx | XX | DD-MMM-YYYY | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | XXXX | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# Listing 16.2.2.2. Listing of Patient Exacerbation (Part 2)

| Patient | Patient visit the emergency room | Number of | Patient Hospitalizations | ICU | General | Patient visit to clinic | Visit | No. of Emergency |
|---|---|---|---|---|---|---|---|---|
| No | due to this Exacerbation | Telephone Call | due to this Exacerbation | (Days) | ward (Days) | as out-patient | (days) | Room Visit (days) |
| XX-XXX | Yes/No | Xx | Yes/No | Xx | Xx | Yes/No | Xx | Yes/No |
| XX-XXX | Yes/No | XX | Yes/No | XX | xx | Yes/No | XX | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# Listing 16.2.2.3. Listing of Patient Exacerbation (Part 3)

| Patient No | Oral/Inhaled Corticosteroids taken for the<br>Exacerbation | Patient intubated for this<br>Exacerbation | Exacerbation medication other than<br>oral/Inhaled corticosteroids taken |
|---|---|---|---|
| XX-XXX | Yes/No | Yes/No | Yes/No |
| XX-XXX | Yes/No | Yes/No | Yes/No |
| XX-XXX | Yes/No | Yes/No | Yes/No |
| XX-XXX | Yes/No | Yes/No | Yes/No |
| XX-XXX | Yes/No | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.2.3. Listing of Patient Blood Eosinophils count

| Patient | | Blood Sample | Date and Time of Blood | | | | Reference | | If Abnormal |
|---|---|---|---|---|---|---|---|---|---|
| No | Visit | Collected | Sample Collected | Parameter | Result | Unit | Range | Assessment | CS |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | Xxxx | Xxxx | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | xxxx | xxxx | xxxx | xxxx | Normal/Abnormal | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.2.4. Listing of Overall Investigators Assessment

| Patient No | Visit | Overall Investigators Assessment performed | If Yes |
|---|---|---|---|
| XX-XXX | XXXX | Yes/No | Well controlled/Partly controlled/Uncontrolled |
| XX-XXX | xxxx | Yes/No | Well controlled/Partly controlled/Uncontrolled |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# Listing 16.3.1.1. Listing of Patient Adverse Event Assessment

| | | Patient Experience any adverse | Patient Experience any new adverse event or change in |
|---|---|---|---|
| Patient No | Visit | event since ICF obtained | existing adverse event since ICF obtained |
| xx-xxx | XXXX | Yes/No | Yes/No |
| xx-xxx | XXXX | Yes/No | Yes/No |
| xx-xxx | XXXX | Yes/No | Yes/No |
| xx-xxx | xxxx | Yes/No | Yes/No |
| xx-xxx | XXXX | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# Listing 16.3.1.2. Listing of Patient Adverse Events

| | Patient | | | | | | Investigators causality | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | Experience any | Seq. | Event | Start Date/Stop | | | rating against the | Action | Patient | Treatment | | |
| No | Adverse Event | No. | Description | Date | Ongoing | Intensity | <b>Investigational Product</b> | taken | Withdrawn | taken | Outcome | SAE |
| | | | | DD-MMM-YYYY/ | | | | | | | | |
| XX-XXX | Yes/No | Xx | Xxxx | DD-MMM-YYYY | Xxxx | Xxxx | Yes/No | Xxxx | Yes/No | Xxxx | Xxxx | Yes/No |
| | | | | DD-MMM-YYYY/ | | | | | | | | |
| XX-XXX | Yes/No | XX | Xxxx | DD-MMM-YYYY | Xxxx | Xxxx | Yes/No | Xxxx | Yes/No | Xxxx | Xxxx | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# Listing 16.3.2.1. Listing of Patient Serious Adverse Events (Part 1)

| | | | | | Date of Investigator | Patient | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| <b>Patient</b> | | | | Date of AE met | became aware of | Hospitalized | Date of | Date of | Seriousness | Date of Event |
| No | Age | Gender | SAE term | criteria for SAE | Serious AE | due to SAE | Hospitalized | Discharge | Criteria | Onset |
| XX-XXX | Xx | Xx | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY |
| XX-XXX | XX | XX | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# Listing 16.3.2.2. Listing of Patient Serious Adverse Events (Part 2)

| Patient | <b>,</b> | | | Recovered with | Probable Cause | Autopsy | |
|---|---|---|---|---|---|---|---|
| No | relation to study Procedure | relation to other medication | Outcome | sequelae date | of Death | Performed | Date of Autopsy |
| XX-XXX | Yes/No | Yes/No | Xxxx | DD-MMM-YYYY | XXXX | Yes/No | DD-MMM-YYYY |
| XX-XXX | Yes/No | Yes/No | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY |
| XX-XXX | Yes/No | Yes/No | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY |
| xx-xxx | Yes/No | Yes/No | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY |
| XX-XXX | Yes/No | Yes/No | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Applysis Plan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.3.3.1. Listing of Patient Haematology Parameters

| | | Blood Sample | Date and Time of Blood | | | | Reference | | If Abnormal |
|---|---|---|---|---|---|---|---|---|---|
| Patient No | Visit | Collected | sample | Parameter | Result | Unit | Range | Clinical Significance | CS/NCS |
| xx-xxx | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | XXXX |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | XXXX |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | xxxx |
| xx-xxx | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | xxxx | Normal / Abnormal | xxxx |
| xx-xxx | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Applysis Plan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

# Listing 16.3.3.2. Listing of Patient Biochemistry Parameters

| | | Blood Sample | Date and Time of Blood | | | | Reference | | If Abnormal |
|---|---|---|---|---|---|---|---|---|---|
| Patient No | Visit | Collected | sample | Parameter | Result | Unit | Range | Clinical Significance | CS/NCS |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | xxxx | Normal / Abnormal | Xxxx |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | Xxxx |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | Xxxx |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | xxxx | XXXX | XXXX | Normal / Abnormal | Xxxx |
| xx-xxx | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | xxxx | Normal / Abnormal | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Blan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.3.3.3. Listing of Patient Urinalysis Parameters

| | | Blood Sample | Date and Time of Urine | | | | Reference | | If Abnormal |
|---|---|---|---|---|---|---|---|---|---|
| Patient No | Visit | Collected | sample | Parameter | Result | Unit | Range | Clinical Significance | CS/NCS |
| xx-xxx | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | Xxxx |
| xx-xxx | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | XXXX |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | XXXX |
| xx-xxx | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | XXXX |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | Normal / Abnormal | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.3.3.4. Listing of Patient Serum Pregnancy Test

| Patient No | Visit | Serum Pregnancy test performed | Date and Time of Assessment | Result |
|---|---|---|---|---|
| XX-XXX | XX-XXX | Yes/No | DD-MMM-YYYY/HH:MM | Positive/Negative |
| XX-XXX | xx-xxx | Yes/No | DD-MMM-YYYY/HH:MM | Positive/Negative |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.4. Listing of Patient Vital Signs

| | | | | | | | | If Abnormal |
|---|---|---|---|---|---|---|---|---|
| Patient No | Visit | Vital signs collected | If No, Specify reason | Parameter | Result | Unit | Assessment | CS/NCS |
| XX-XXX | XXXX | Yes/No | Xxxx | Xxxx | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| XX-XXX | XXXX | Yes/No | Xxxx | Xxxx | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| XX-XXX | XXXX | Yes/No | Xxxx | Xxxx | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| XX-XXX | xxxx | Yes/No | Xxxx | Xxxx | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | xxxx | XXXX | XXXX | Normal/Abnormal | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.5. Listing of Patient Electrocardiogram (ECG)

| | | ECG | If No, Specify | | | | | If Abnormal |
|---|---|---|---|---|---|---|---|---|
| Patient No | Visit | Performed | reason | Parameter | Result | Unit | Assessment | CS/NCS |
| xx-xxx | xxxx | Yes/No | Xxxx | Xxxx | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| XX-XXX | xxxx | Yes/No | Xxxx | Xxxx | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| XX-XXX | xxxx | Yes/No | Xxxx | Xxxx | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| xx-xxx | xxxx | Yes/No | Xxxx | Xxxx | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| xx-xxx | xxxx | Yes/No | xxxx | XXXX | xxxx | Xxxx | Normal/Abnormal | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.6. Listing of Patient Targeted Physical Examination

| Patient | | Physical Examination | If No, Specify | Date of Physical | Seq. | | | If Abnormal |
|---|---|---|---|---|---|---|---|---|
| No | Visit | performed | reason | Examination | No | System | Assessment | CS/NCS |
| XX-XXX | XXXX | Yes/No | Xxxx | DD-MMM-YYYY | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| XX-XXX | XXXX | Yes/No | Xxxx | DD-MMM-YYYY | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| XX-XXX | XXXX | Yes/No | Xxxx | DD-MMM-YYYY | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| xx-xxx | XXXX | Yes/No | Xxxx | DD-MMM-YYYY | Xxxx | Xxxx | Normal/Abnormal | Xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY | XXXX | XXXX | Normal/Abnormal | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.7. Listing of Patient Urinalysis Pregnancy test

| Patient No | Visit | Urine Pregnancy Test performed | Date and Time of Assessment | Result |
|---|---|---|---|---|
| XX-XXX | Xxxx | Yes/No | DD-MMM-YYYY/HH:MM | Positive/Negative |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | Positive/Negative |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | Positive/Negative |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | Positive/Negative |
| XX-XXX | xxxx | Yes/No | DD-MMM-YYYY/HH:MM | Positive/Negative |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.8. Listing of Patient Pregnancy Form

| | | Date of Last | Date of | Outcome | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| <b>Patient</b> | Date Pregnancy | Menstrual | Estimated | of | | Pregnancy | Elective | Spontaneous/ | Ectopic |
| No | was confirmed | Period | delivery | Pregnancy | Live Birth Date | Status | abortion Date | misses Date | abortion Date |
| XX-XXX | DD-MMM-YYYY | DD-MMM-YYYY | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY | DD-MMM-YYYY | DD-MMM-YYYY |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.9.1. Listing of Patient Concomitant Medication

| Patient No | Visit | Patient have any other concomitant medication during visit | Aby changes in concomitant or taking new medication since last visit |
|---|---|---|---|
| xx-xxx | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.9.2. Listing of Patient Prior and Concomitant Medication

| | Patient receive any | Seq | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | Prior or concomitant | | Medication | Start Date/Stop | | | Indication | Dosage | | | | |
| No | medications | No. | Name | Date | Ongoing | Indication | Description | Form | Dose | Unit | Route | Frequency |
| | | | | DD-MMM-YYYY/ | | | | | | | | |
| XX-XXX | Yes/No | Xx | Xxxx | DD-MMM-YYYY | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| | | | | DD-MMM-YYYY/ | | | | | | | | |
| XX-XXX | Yes/No | Xx | Xxxx | DD-MMM-YYYY | xxxx | xxxx | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| | | | | DD-MMM-YYYY/ | | | | | | | | |
| XX-XXX | Yes/No | Xx | Xxxx | DD-MMM-YYYY | xxxx | xxxx | XXXX | xxxx | XXXX | XXXX | XXXX | XXXX |
| | | | | DD-MMM-YYYY/ | | | | | | | | |
| XX-XXX | Yes/No | Xx | Xxxx | DD-MMM-YYYY | xxxx | xxxx | XXXX | xxxx | XXXX | XXXX | XXXX | XXXX |
| | | | | DD-MMM-YYYY/ | | | | | | | | |
| XX-XXX | Yes/No | XX | Xxxx | DD-MMM-YYYY | XXXX | xxxx | XXXX | xxxx | XXXX | XXXX | XXXX | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Figure 14.2.1. Figure of Time to first Asthma Exacerbation



Programmer Note: Kaplan-Meier Curve format will change.; X-axis= Time (Days) and y- axis=Probability



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Figure 14.2.2. Figure of Number of Exacerbation



Programmer Note: X-axis= Time point and y- axis= No. of Excerbations



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Figure 14.2.3. Figure of Mean of Exacerbation



Programmer Note: X-axis= Time point and y- axis= Mean of Excerbations